CLINICAL TRIAL: NCT04761224
Title: Impact of Intraoperative Instillation of Normothermal Saline on the Prevention of Intraoperative Hypothermia and Perioperative Morbidity of Prostatic Enucleation With Holmium Laser: a Prospective Randomized Controlled Study
Brief Title: Impact of Intraoperative Instillation of Normothermal Saline on the Prevention of Intraoperative Hypothermia and Perioperative Morbidity of Prostatic Enucleation With Holmium Laser
Acronym: THERMHOLEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: THERMHOLEP
Record Dates: First submitted 2021-02-08; First posted 2021-02-18 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Prostatic Hypertrophy
Keywords: normothermal solution; enucleation; hypothermia
MeSH Terms: conditions — Prostatic Hyperplasia; Hypothermia

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The surgeon cannot be blind to the treatment group. On the other hand, the treatment group will be masked for all the participants (doctors and nurses) in charge of collecting the judgement criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): heated blanket + unheated NaCL instillation (operating room ambient temperature: around 17°C).
- Heated group (Experimental): heating blanket + instillation of NaCl at 38-39°C by Fluido® Irrigation fluid heating system
  Interventions: Device: Fluido® Irrigation Fluid Heater System

INTERVENTIONS:
Device: Fluido® Irrigation Fluid Heater System — Patients in the "Heated" group will benefit from intraoperative warming by means of NaCl bags instilled using the Fluido® Irrigation warming cassette and with the use of specific instillation tubing (SEBAC laboratory, Set URO Fluido® Irrigation): this device allows continuous and precise heating of the solution with an instillation temperature of 38-39°C.
  Arms: Heated group

SUMMARY:
For the treatment of benign prostatic hyperplasia (BPH), 2 types of endoscopic surgery are currently performed: transurethral prostate resection (TPR), the reference surgery, and laser prostatic enucleation (LPE). These procedures can be performed under general anesthesia, or local anesthesia, such as spinal anesthesia. The EPL or RTUP procedure requires the instillation of continuous intra-vesical fluids throughout the procedure. These 3L bags are often kept at the ambient temperature of the operating room (around 17°C): the temperature of the instilled solution is therefore much lower than the average body temperature of the patient (37°C). Thus, and by heat exchange, it often results in per and postoperative hypothermia, which is all the more frequent and profound the longer the duration of the operation.

In spite of the usual procedures of warming by heating blanket, the prevalence of hypothermia, defined as a body temperature < 36°C, is 53.5% during surgical procedures. This hypothermia is all the more frequent and profound the older the patient is and the longer the duration of anesthesia.

Several studies have shown that hypothermia is particularly frequent during abdomino-pelvic surgery, notably due to pathophysiological phenomena induced by anesthetic procedures. Indeed, general anesthesia, or major locoregional anesthesia, disrupts the thermoregulation center upon anesthetic induction, with alteration of peripheral vasoconstriction and tremor capacity, leading to a rapid redistribution of body heat from the center to the periphery. Through exchanges with the environment, this results in a rapid linear decrease in central body temperature that exceeds the metabolic energy produced.

However, anesthetic procedures are not the only cause of hypothermic intraoperative phenomena. It has been shown that the decrease in body temperature associated with most genitourinary endoscopic procedures is multifactorial, taking into account the patient's body mass, the volume of fluids instilled, and the type and duration of the operation.

DETAILED DESCRIPTION:
Even moderate hypothermia (body temperature between 34-36°C) would contribute significantly to the increase in postoperative morbidity and mortality. Indeed, it would significantly increase blood loss (16%) with an increased relative risk of transfusion (22%) by altering platelet aggregation and coagulation cascade enzyme function. It would also be responsible for an increase in the risk of infection and length of hospitalization, alteration of drug metabolism (accumulation of serum curare and delayed awakening) and a decrease in postoperative tremors, which can lead to severe cardiovascular complications (myocardial infarction, heart rhythm disorder, etc.).

Due to the instillation of hypothermic solution, perioperative hypothermia is frequent in endoscopic surgery (arthroscopy, abdominal laparoscopy, endoscopic prostate resection...), in the order of 48% to 64%. Several studies have evaluated the impact of pre- and intraoperative warming procedures. Thus, intraoperative external body heating would decrease the risk of hypothermia and its complications during RTUP. Similarly, the use of heated intravenous fluids has been shown to decrease the depth of hypothermia (+0.5°C) during endoscopic surgery and RTUP.

Several authors have examined the warming of IV bags instilled during RTUP procedures, the reference endoscopic surgery for BPH management. Pit et al. have shown a significant increase in postoperative body temperature in patients who underwent RTUP with isothermal solutions compared to the group undergoing a standard procedure (- 0.74°C versus -1.71°C, p < 0.05). These results were corroborated by the study by Singh et al. but none of these studies evaluated the impact of these measures on postoperative morbidity nor showed a statistical impact on intraoperative blood loss.

Holmium Laser Enucleation of the Prostate (HoLEP) is an endoscopic surgical technique that was first described by Gilling in New Zealand in 1998, and is indicated since 2013 as an alternative to RTUP for the management of symptomatic BPH. It requires continuous intravesical instillation of saline throughout the procedure. The complication rate in the 30 days postoperatively is 19 to 25%, and this risk increases with the duration of the surgery, which in turn is directly correlated to the volume of prostate to be enucleated.

Currently, only one study has studied the consequences of hypothermia during EPL procedures: the authors have shown that external body preheating to a temperature of 41°C, in the induction room, would increase the intraoperative temperature by + 0.2°C on average, and would therefore reduce the incidence of tremors during EPL performed under spinal anesthesia. On the other hand, the investigators did not find any study on the impact of warming of solutes during HoLEP, either on the immediate postoperative incidence in the post-operative monitoring room (SSPI) or on morbidity in the post-operative period.

This study thus consists in analyzing, in a prospective manner, the effect of warming of the solutes instilled during HoLEP on the post-operative morbidity of patients. To the investigators' knowledge, this is the first study of this type in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Male patient whose age is ≥ 18 years old
* Patient eligible for holmium laser prostate enucleation
* Patient affiliated to a social security system
* Francophone patient
* Patient who has given free, informed and written consent

Exclusion Criteria:

* Patient already included in a Type 1 Intervention Research Protocol (RIPH1)
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of warming patients by intravesical instillation of warmed intravesical fluid using the Fluido® Irrigation device, by assessing the rate of hypothermic patients on arrival in post-procedural follow-up care. | Day 1
  Rate of hypothermic patients (< 36°C) on arrival in post-procedural follow-up care.

SECONDARY OUTCOMES:
Evaluate the variation of body temperature intraoperatively | Day 1
  Temperature difference between entry into the operating room and arrival in post-operative follow-up care (in °C)
Duration of general anesthesia | Day 1
  Time between anesthetic induction and extubation (in min)
Complications rate within 30 days postoperatively | Day 30
  Complications according to Clavien- Dindo (%)
Rate of complications in the 30 days postoperatively according to preoperative prostate weight (< 100g, ≥ 100g but ≤ 200g, > 200g) | Day 30
  Complications according to Clavien- Dindo (%)
Rate of serious complications within 30 days postoperatively | Day 30
  Complications Clavien-Dindo ≥ III (%)
ECG modifications induced by hypothermia | Day 30
  Rate of ECG changes in post-procedural follow-up care (%)
Serum troponin modifications induced by hypothermia | Day 30
  Change in serum troponin between Day 0 and Day 1 (ng/L)
Hb loss > 2g/dL postoperatively | Day 30
Transfusion within 30 days postoperatively | Day 30
Unblocking at the patient's bedside | Day 30
Surgical resection for unblocking | Day 30
Re - admission within 30 days postoperatively for macroscopic hematuria | Day 30
Duration of bladder catheterization | Day 1
  Number of days of bladder catheterization
Evaluation of the length of hospital stay | An average of 2 days
  Number of days in hospital
International Prostate Symptom Score (IPSS score) | 3 months
  0 - 7 = mild 8 - 19 = moderate 20 - 35 = severe
International Prostate Symptom Score (IPSS score) | 12 months
  0 - 7 = mild 8 - 19 = moderate 20 - 35 = severe
Functional evaluation | 3 months
  Quality of Life score (QoL score)
  0 = very satisfied 6 = very bored
Functional evaluation | 12 months
  Quality of Life score (QoL score)
  0 = very satisfied 6 = very bored
5-item version of the International Index of Erectile Function ( IIEF-5) | 3 months
  1 - 4 = Not interpretable 5 - 10 = Severe erectile dysfunction 11 - 15 = Moderate erectile dysfunction 16 - 20 = Mild erectile dysfunction 21 - 25 = Normal erectile function
5-item version of the International Index of Erectile Function ( IIEF-5) | 12 months
  1 - 4 = Not interpretable 5 - 10 = Severe erectile dysfunction 11 - 15 = Moderate erectile dysfunction 16 - 20 = Mild erectile dysfunction 21 - 25 = Normal erectile function

CONTACTS AND LOCATIONS:
Overall Officials: Constance MICHEL, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France